CLINICAL TRIAL: NCT06482541
Title: 1-Year Double-Blind Placebo-Controlled Study To EVALUATE THE EFFECT OF AGE ZERO™ EXOSOMES ON HAIR REGROWTH IN HEALTHY MEN AND WOMEN WITH ANDROGENETIC ALOPECIA
Brief Title: Efficacy and Safety Of AGE ZERO™ EXOSOMES To Treat Men and Women With Androgenetic Alopecia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Levit Dermatology (Other)
Collaborators: ResilielleTM Age ZeroTM Exosomes (Unknown); Dorisca Research Consulting, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-06-001
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Androgenetic Alopecia
Keywords: exosomes; Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Participants will act as their own control. Each participant will get exosome treatment on one half of the treatment area and placebo on the other half of the treatment area. The treatment area will be two rectangles each measuring 4cm on the sagittal plane by 2cm on the coronal plane on the scalp vertex. One rectangle will be 2.0 mm left of the midline of the scalp and another will be 2.0 mm right of the midline of the scalp. Participants in the 5 billion exosome group will receive 5 billion WJMSC-exosome treatment on one side of the treatment area and an equivalent volume of saline on the other side of the treatment area. Participants in the 50 billion exosome group will receive 5 billion WJMSC-exosome treatment on one side of the treatment area and an equivalent volume of placebo on the other side of the treatment area.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5 billion exosome group (Experimental): This arm receives 5 billion WJMSC-exosome treatment on one side of the aforementioned treatment area and an equivalent volume of placebo on the contralateral half of the treatment area.
  Interventions: Combination Product: 5 billion exosomes and saline solution microneedling
- 50 billion exosome group (Experimental): This arm receives 50 billion WJMSC-exosome treatment on one half of the aforementioned treatment area and an equivalent volume of placebo on the contralateral half of the treatment area.
  Interventions: Combination Product: 50 billion exosomes and saline solution microneedling

INTERVENTIONS:
Combination Product: 5 billion exosomes and saline solution microneedling — Participants will receive 5 billion WJMSC-exosome topical application on one half of the treatment area and an equivalent volume of saline solution on the contralateral half of the treatment area. Microneedling at a depth of .5mm on the entire treatment area will immediately follow the exosome and saline application. Participants will also receive 4 permanent microdot tattoos on the aforementioned locations.
  Arms: 5 billion exosome group
Combination Product: 50 billion exosomes and saline solution microneedling — Participants will receive 50 billion WJMSC-exosome topical application on one half of the treatment area and an equivalent volume of saline solution on the contralateral half of the treatment area. Microneedling at a depth of .5mm on the entire treatment area will immediately follow the exosome and saline application. Participants will also receive 4 permanent microdot tattoos on the aforementioned locations.
  Arms: 50 billion exosome group

SUMMARY:
The purpose of this study is to determine whether Wharton's Jelly mesenchymal stem cell-derived exosome microneedling on the scalp is an effective treatment for Androgenetic Alopecia (pattern hair loss).

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants who give written consent and meet the later discussed inclusion criteria and don't fall under the exclusion criteria will be enrolled in the study.

The investigators will conduct a double-blind placebo-controlled study to test whether Wharton's Jelly Mesenchymal Stem Cell-derived Exosome (WJMSC-exosome) application with microneedling is an effective treatment for Androgenetic Alopecia. Participants will be broken down into a 5 billion exosome group vs. saline group and a 50 billion exosome vs. saline group.

Treatment will be applied to the following treatment area: two rectangles on the scalp vertex each measuring 4cm on the sagittal plane by 2cm on the coronal plane. One rectangle will be 2.0 mm left of the midline of the scalp and another will be 2.0 mm right of the midline of the scalp. Each treatment area will be divided into an anterior and posterior half with 1 permanent microdot tattoo in the middle (4 tattoos in total). The microdot tattoo (composed of Iron Oxide, Glycerol, Alcohol, and distilled Water and Red - D&C Red #30, Glycerol, Alcohol and distilled water) will allow HairMatrix® by Canfield, an AI-driven hair consultation device, to accurately and reproducibly access changes in hair growth in the treatment areas.

Participants in the 5 billion exosome group will receive topical applications of 5 billion WJMSC-exosomes on one side of the treatment area and an equal volume of placebo (an identically-looking saline solution) application on the opposite side of the treatment area.

The 50 billion exosome group will receive topical applications of 50 billion WJMSC-exosomes on one side of the treatment area and an equal volume of placebo application on the opposite side of the treatment area.

Immediately after topical application, all participants will receive microneedling at a depth of .5 mm on the entire treatment area.

Treatment will be administered in 4 sessions, monthly for the first three months and for a 4th time 4 months after the third session.

The study will go on for 12 months from the date of the first treatment. Participant's changes in hair growth (hair count, hair thickness, and hair color) and adverse events will be evaluated and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Participant is experiencing hair loss and is diagnosed with Androgenetic Alopecia.

Exclusion Criteria:

* Patients cannot have taken any medications, therapies, or treatment modalities of any kind to treat hair loss in the last six months.
* Patients cannot have open wounds, eczema, or psoriatic plaques on the treatment area of the scalp.
* Patients who are undergoing or have undergone chemotherapy and or radiation therapy within the past 6 months
* Patients with a history of an autoimmune bullous disorder (having auto-antibodies to Dsg-1 or Dsg-3)
* Patients who are currently immunocompromised or have a low white count making patients prone to infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Hair count | Evaluated on monthly visits for a year
  Evaluated by HairMatrix® by Canfield, an AI-driven hair consultation device
Hair thickness | Evaluated on monthly visits for a year
  Evaluated by HairMatrix® by Canfield, an AI-driven hair consultation device
Hair color | Evaluated on monthly visits for a year
  Evaluated by HairMatrix® by Canfield, an AI-driven hair consultation device

SECONDARY OUTCOMES:
Adverse events | Participants will self-report adverse events during monthly visits for the entire 1-year duration
  Patients will self-report adverse events on a questionnaire on a scale of 1-10, with 1 being minimal discomfort and 10 being worst discomfort ever experienced.
Self-reported hair changes | Patients will self-report on questionnaire during monthly visits for the entire 1-year duration
  Patients will self-report impressions of hair growth changes on each treatment area on a scale of -10 to 10, with -10 being extreme worsening of hair loss and 10 being extreme regrowth. Patients will scale impressions of hair thickness, hair density, hair color, hair growth speed, hair texture, and overall satisfaction with therapy applied to each treatment area.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal K Levit, M.D., Principal Investigator — Owner and chief physician
Locations (1):
- Levit Dermatology, Brooklyn, New York, United States